CLINICAL TRIAL: NCT01704755
Title: A Randomized, Open-Label Study to Evaluate the Safety and Efficacy of ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 Coadministered With Ribavirin (RBV) in Adults With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection and Cirrhosis (TURQUOISE-II)
Brief Title: A Study to Evaluate the Safety and Efficacy of ABT-450/Ritonavir/ABT-267; (ABT-267 Also Known as Ombitasvir) and ABT-333 (Also Known as Dasabuvir) Coadministered With Ribavirin (RBV) in Hepatitis C Virus (HCV) Genotype 1-infected Adults With Compensated Cirrhosis
Acronym: TURQUOISE-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13-099; 2012-003088-23 (EudraCT Number)
Record Dates: First submitted 2012-09-28; First posted 2012-10-11 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C Infection; Compensated Cirrhosis
Keywords: Cirrhosis; Hepatitis C; Child Pugh A; Compensated Cirrhosis; Hepatitis C Genotype 1; Cirrhotic; Chronic Hepatitis C; Hepatitis C Virus; ombitasvir; paritaprevir; dasabuvir; Interferon-Free; Viekira Pak
MeSH Terms: conditions — Fibrosis; Hepatitis C; Hepatitis C, Chronic | interventions — dasabuvir; Viekira Pak; paritaprevir; ombitasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABT-450/r/ABT-267 and ABT-333, plus RBV for 12 weeks (Experimental): ABT-450/r/ABT-267 (150/100/25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based ribavirin (RBV; 1,000 mg/day if <75 kg or 1,200 mg/day if ≥75 kg, divided twice daily) for 12 weeks
  Interventions: Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)
- ABT-450/r/ABT-267 and ABT-333, plus RBV for 24 weeks (Experimental): ABT-450/r/ABT-267 (150/100/25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based ribavirin (RBV; 1,000 mg/day if <75 kg or 1,200 mg/day if ≥75 kg, divided twice daily) for 24 weeks
  Interventions: Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: ABT-450/r/ABT-267, ABT-333 — Tablet; ABT-450 coformulated with ritonavir and ABT-267; ABT-333 tablet
  Other Names: Viekira Pak; ABT-450 also known as paritaprevir; ABT-267 also known as ombitasvir; ABT-333 also known as dasabuvir
Drug: Ribavirin (RBV) — Capsule

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ABT-450/ritonavir/ABT-267 (ABT-450/r/ABT-267; ABT-450 also known as paritaprevir; ABT-267 also known as ombitasvir) and ABT-333 (also known as dasabuvir) coadministered with ribavirin (RBV) in hepatitis C virus (HCV) genotype 1-infected adults with compensated cirrhosis.

DETAILED DESCRIPTION:
During the treatment period of the study, participants received treatment with ABT-450/ritonavir/ABT-267 and ABT-333 coadministered with RBV for either 12 or 24 weeks. Upon completing the treatment period or premature discontinuation of the treatment period, participants entered a 48-week post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Females must be practicing specific forms of birth control on study treatment, or be post-menopausal for more than 2 years or surgically sterile
* Male or female between 18 and 70 years, inclusive, at time of Screening.
* Chronic HCV-infection prior to study enrollment.
* Screening laboratory result indicating HCV genotype 1-infection.
* Compensated cirrhosis defined as a Child-Pugh Score of less than or equal to 6 at Screening
* Subject has plasma HCV RNA level greater than 10,000 IU/mL at Screening.

Exclusion Criteria:

* Significant liver disease with any cause other than HCV as the primary cause
* Positive test result for Hepatitis B surface antigen (HBsAg) or anti-Human Immunodeficiency virus antibody (HIV Ab) at screening.
* Prior therapy with direct acting antiviral agents for the treatment of HCV, including telaprevir and boceprevir.
* Any current or past clinical evidence of Child-Pugh B or C Classification or clinical history of liver decompensation including ascites (noted on physical exam), variceal bleeding or hepatic encephalopathy.
* A positive screening ultrasound for hepatocellular carcinoma (HCC) confirmed with a subsequent CT Scan or MRI during the screening period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Trinh, MD, Study Director — AbbVie

REFERENCES:
- [Background] Poordad F, Hezode C, Trinh R, Kowdley KV, Zeuzem S, Agarwal K, Shiffman ML, Wedemeyer H, Berg T, Yoshida EM, Forns X, Lovell SS, Da Silva-Tillmann B, Collins CA, Campbell AL, Podsadecki T, Bernstein B. ABT-450/r-ombitasvir and dasabuvir with ribavirin for hepatitis C with cirrhosis. N Engl J Med. 2014 May 22;370(21):1973-82. doi: 10.1056/NEJMoa1402869. Epub 2014 Apr 11. PMID 24725237
- [Derived] Feld JJ, Bernstein DE, Younes Z, Vlierberghe HV, Larsen L, Tatsch F, Ferenci P. Ribavirin dose management in HCV patients receiving ombitasvir/paritaprevir/ritonavir and dasabuvir with ribavirin. Liver Int. 2018 Sep;38(9):1571-1575. doi: 10.1111/liv.13708. Epub 2018 Mar 14. PMID 29377566
- [Derived] Forns X, Poordad F, Pedrosa M, Berenguer M, Wedemeyer H, Ferenci P, Shiffman ML, Fried MW, Lovell S, Trinh R, Lopez-Talavera JC, Everson G. Ombitasvir/paritaprevir/r, dasabuvir and ribavirin for cirrhotic HCV patients with thrombocytopaenia and hypoalbuminaemia. Liver Int. 2015 Nov;35(11):2358-62. doi: 10.1111/liv.12931. Epub 2015 Sep 6. PMID 26248955
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the 12-week treatment group, one participant withdrew from the study before receiving study drug.
Period: Overall Study
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks
Started | 208 | 172
Completed Study Drug | 204 | 163
Completed | 196 | 165
Not Completed | 12 | 7
Not completed — Adverse Event | 4 | 1
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrew consent | 1 | 1
Not completed — Other (not specified) | 3 | 1
Not completed — Withdrew consent and personal issues | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks | Total
Number analyzed (Participants) | 208 | 172 | 380
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (7.01) | 56.5 (7.87) | 56.8 (7.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 51 | 113
  Male | 146 | 121 | 267

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks
Number analyzed (Participants) | 208 | 172
Percentage of participants | 91.8 | 96.5
Statistical Analysis 1: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks; The study planned to enroll 380 subjects to a 12- or 24-week treatment arm. The primary efficacy endpoint (SVR12) was assessed for each arm. With a total sample size of 380 and assuming that 68% of the subjects in each arm would achieve SVR12, the study had greater than 90% power to demonstrate non-inferiority and superiority with a 2-sided 97.5% lower confidence bound greater than 43% and 54%, respectively, based on the normal approximation of a single binomial proportion; Test type: Non-Inferiority or Equivalence — The noninferiority of the rate of sustained virologic response for the ABT-450/r/ABT-333 plus ribavirin 12-week treatment group as compared with the historical rate for telaprevir plus peginterferon-ribavirin. The lower confidence bound of the 2-sided 97.5% CI for the percentage of participants with sustained virologic response at 12 weeks after treatment must have exceeded 43% to achieve noninferiority; Percentage of Participants = 91.8, 97.5% CI 2-sided [87.6 to 96.1]
Statistical Analysis 2: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks; The primary efficacy endpoints were the SVR12 rates in each arm. The overall 2-sided significance level of 0.05 was split between the arms using a Bonferroni correction of 0.025. A 2-sided 97.5% CI of the SVR12 rate per arm was computed using the normal approximation to the binomial distribution. A gatekeeping testing procedure was used to control the Type I error rate at 0.05, and the primary endpoints for Arm A were tested separately from Arm B in a pre-specified order; Test type: Non-Inferiority or Equivalence — The superiority of the rate of sustained virologic response for the ABT-450/r/ABT-333 plus ribavirin 12-week treatment group as compared with the historical rate for telaprevir plus peginterferon-ribavirin. The lower confidence bound of the 2-sided 97.5% CI for the percentage of participants with sustained virologic response at 12 weeks after treatment must have exceeded 54% to achieve superiority; Percentage of Participants = 91.8, 97.5% CI 2-sided [87.6 to 96.1]
Statistical Analysis 3: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks; Test type: Non-Inferiority or Equivalence — The noninferiority of the rate of sustained virologic response for the ABT-450/r/ABT-333 plus ribavirin 24-week treatment group as compared with the historical rate for telaprevir plus peginterferon-ribavirin. The lower confidence bound of the 2-sided 97.5% CI for the percentage of participants with sustained virologic response at 12 weeks after treatment must have exceeded 43% to achieve noninferiority; Percentage of Participants = 96.5, 97.5% CI 2-sided [93.4 to 99.7]
Statistical Analysis 4: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks; Test type: Non-Inferiority or Equivalence — The superiority of the rate of sustained virologic response for the ABT-450/r/ABT-333 plus ribavirin 24-week treatment group as compared with the historical rate for telaprevir plus peginterferon-ribavirin. The lower confidence bound of the 2-sided 97.5% CI for the percentage of participants with sustained virologic response at 12 weeks after treatment must have exceeded 54% to achieve superiority; Percentage of Participants = 96.5, 97.5% CI 2-sided [93.4 to 99.7]

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment in the 24-week Arm Compared to the 12-week Arm
Description: A sustained virologic response is defined as plasma Hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (< LLOQ) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks
Number analyzed (Participants) | 208 | 172
Percentage of participants | 91.8 | 96.5
Statistical Analysis 1: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks vs ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks; To test the hypothesis that the percentages of participants who achieved sustained virologic response 12 weeks after treatment was different between the two treatment groups, the percentages were compared using a logistic regression model with treatment group, baseline log(subscript)10(subscript) HCV RNA level, HCV subgenotype (1a, non-1a), IL28B genotype (CC, non CC), and peginterferon-ribavirin treatment history (treatment-naïve or treatment-experienced) as predictors; Test type: Superiority or Other; p = 0.051, Regression, Logistic

3. Secondary Outcome: Percentage of Participants in Each Arm With On-treatment Virologic Failure During the Treatment Period
Description: Virologic failure during treatment was defined as rebound (confirmed HCV RNA greater than or equal to the lower limit of quantitation [≥ LLOQ] after HCV RNA < LLOQ during treatment, or confirmed increase from the lowest value post baseline in HCV RNA [2 consecutive HCV RNA measurements > 1 log(subscript)10(subscript) IU/mL above the lowest value post baseline] at any time point during treatment), or fail to suppress (HCV RNA ≥ LLOQ persistently during treatment with at least 6 weeks [≥ 36 days] of treatment).
Time Frame: Baseline (Day 1), and Treatment Weeks 1, 2, 4, 6, 8, 10, 12, 16, 20, and 24
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks
Number analyzed (Participants) | 208 | 172
Percentage of participants | 0.5 [0.0 to 1.4] | 1.7 [0.0 to 3.7]

4. Secondary Outcome: Percentage of Participants With Virologic Relapse After Treatment
Description: Participants were considered to have virologic relapse after treatment if they had confirmed quantifiable plasma Hepatitis C virus ribonucleic acid (HCV RNA) ≥ lower limit of quantification (LLOQ) between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA < LLOQ at the end of treatment.
Time Frame: within 12 weeks after the last dose of study drug
Population: All randomized participants who received at least 1 dose of study drug with HCV RNA < LLOQ at the final treatment visit who completed treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks
Number analyzed (Participants) | 203 | 164
Percentage of participants | 5.9 [2.7 to 9.2] | 0.6 [0.0 to 1.8]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration until 30 days after the last dose, 16 weeks for the 12-week treatment group and 28 weeks for the 24-week treatment group.
Description: Serious adverse events were collected from the time of informed consent until the end of participation in the study (up to 72 weeks).
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks
Serious Adverse Events (participants affected / at risk) | 13/208 | 7/172
Other Adverse Events (participants affected / at risk) | 175/208 | 146/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks (N=208) | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks (N=172)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
MELAENA (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 | 0
CANDIDIASIS (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 1
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 | 0
WOUND (Injury, poisoning and procedural complications) | 1 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 1
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 | 1
MAJOR DEPRESSION (Psychiatric disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 12 Weeks (N=208) | ABT-450/r/ABT-267 and ABT-333, Plus RBV for 24 Weeks (N=172)
ANAEMIA (Blood and lymphatic system disorders) | 15 | 17
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 6 | 9
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 11 | 16
DIARRHOEA (Gastrointestinal disorders) | 30 | 29
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 7 | 10
NAUSEA (Gastrointestinal disorders) | 36 | 35
VOMITING (Gastrointestinal disorders) | 6 | 14
ASTHENIA (General disorders) | 29 | 22
FATIGUE (General disorders) | 68 | 80
IRRITABILITY (General disorders) | 15 | 21
OEDEMA PERIPHERAL (General disorders) | 12 | 10
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 15 | 2
NASOPHARYNGITIS (Infections and infestations) | 13 | 13
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 13
BLOOD BILIRUBIN INCREASED (Investigations) | 12 | 9
DECREASED APPETITE (Metabolism and nutrition disorders) | 12 | 14
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 10 | 14
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 13
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 14 | 14
DIZZINESS (Nervous system disorders) | 18 | 10
HEADACHE (Nervous system disorders) | 58 | 53
MEMORY IMPAIRMENT (Nervous system disorders) | 5 | 12
ANXIETY (Psychiatric disorders) | 15 | 14
DEPRESSION (Psychiatric disorders) | 8 | 12
INSOMNIA (Psychiatric disorders) | 32 | 31
COUGH (Respiratory, thoracic and mediastinal disorders) | 24 | 19
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 12 | 21
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 13 | 11
DRY SKIN (Skin and subcutaneous tissue disorders) | 18 | 11
PRURITUS (Skin and subcutaneous tissue disorders) | 38 | 33
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 10 | 12
RASH (Skin and subcutaneous tissue disorders) | 23 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.